CLINICAL TRIAL: NCT01581658
Title: A Phase I, Open-label, Parallel-group Study to Investigate Pharmacokinetics, Pharmacodynamics and Safety of a Single 25 mg Dose of Empagliflozin in Japanese Type 2 Diabetes Patients With Different Degrees of Renal Impairment in Comparison to Type 2 Diabetes Patients With Normal Renal Function
Brief Title: Renal Impairment Study of Empagliflozin (BI10773) in Japanese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.53
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (4):
- BI10773 medium dose group 1 (Experimental): BI10773 medium dose tablet single dose group 1
  Interventions: Drug: BI10773
- BI10773 medium dose group 2 (Experimental): BI10773 medium dose tablet single dose group 2
  Interventions: Drug: BI10773
- BI10773 Medium dose group 3 (Experimental): BI10773 medium dose tablet single dose group 3
  Interventions: Drug: BI10773
- BI10773 Medium dose group 4 (Experimental): BI10773 medium dose tablet single dose group 4
  Interventions: Drug: BI10773

INTERVENTIONS:
Drug: BI10773 — BI10773 medium dose tablet single dose
  Arms: BI10773 medium dose group 2
Drug: BI10773 — BI10773 medium dose tablet single dose
  Arms: BI10773 Medium dose group 4
Drug: BI10773 — BI10773 medium dose tablet single dose
  Arms: BI10773 medium dose group 1
Drug: BI10773 — BI10773 medium dose tablet single dose
  Arms: BI10773 Medium dose group 3

SUMMARY:
The objective of this study is to assess the effect of the different degrees of renal impairment on the pharmacokinetics, pharmacodynamics and safety of BI10773 following oral administration of high dose BI10773 as a single dose in Japanese patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes patients
* Glycosylated haemoglobin>= 6.1% (Japan Diabetes Society)
* Estimated glomerular filtration rate based on the modification of diet in renal disease-formula at screening , of >= 15 mL/min/1.73m2

Exclusion criteria:

* Any evidence of significant disease (other than renal impairment)
* Moderate and severe concurrent liver function impairment
* Gastrointestinal tract surgery, that might affect absorption and elimination of drugs
* Diseases of the central nervous system (such as epilepsy), psychiatric disorders, or neurological disorders
* Chronic or relevant acute infections
* Participation in another trial with investigational drug administration within 30 days prior to study drug administration or during the trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2012-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.53.001 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka, Japan

REFERENCES:
- [Derived] Sarashina A, Ueki K, Sasaki T, Tanaka Y, Koiwai K, Sakamoto W, Woerle HJ, Salsali A, Broedl UC, Macha S. Effect of renal impairment on the pharmacokinetics, pharmacodynamics, and safety of empagliflozin, a sodium glucose cotransporter 2 inhibitor, in Japanese patients with type 2 diabetes mellitus. Clin Ther. 2014 Nov 1;36(11):1606-15. doi: 10.1016/j.clinthera.2014.08.001. Epub 2014 Sep 5. PMID 25199997

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Renal Function: 25 mg empagliflozin taken as a single dose for patients with normal renal function
- Mild Renal Impairment: 25 mg empagliflozin taken as a single dose for patients with mild renal impairment
- Moderate Renal Impairment: 25 mg empagliflozin taken as a single dose for patients with moderate renal impairment
- Severe Renal Impairment: 25 mg empagliflozin taken as a single dose for patients with severe renal impairment
Period: Overall Study
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (3.1) | 67.5 (4.4) | 65.9 (5.5) | 62.0 (7.9) | 65.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 0 | 2 | 9
  Male | 4 | 5 | 8 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Urinary Glucose Excretion (UGE)
Description: change from baseline in total urinary glucose excretion (UGE) to 24 hours
Time Frame: baseline and 24 hours
Population: Treated patients who had complete urine sample (baseline and 24 hours) for analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 6 | 8 | 7
mg | 74969.3 (4840.68) [64978.6 to 84960.0] | 62577.4 (5751.25) [50707.5 to 74447.4] | 57889.0 (4861.26) [47855.9 to 67922.2] | 23725.1 (5235.06) [12920.5 to 34529.7]

2. Primary Outcome: Area Under the Concentration Time Curve of the Analyte in Plasma
Description: Area under the concentration time curve of the analyte in plasma over the time interval from 0 to infinity
Time Frame: Predose and 20 minutes (min), 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 14h, 24h, 36h 48h, 72h and 96h after drug administration
Population: Treated patients
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
nmol*h/L | 7480 (16.2) | 9630 (15.9) | 10800 (9.55) | 11400 (40.4)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority or Other; ANOVA; The model includes fixed effect for the renal function group; Geometric mean ratio = 128.82, 90% CI 2-sided [105.962 to 156.604]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority or Other; ANOVA; The model includes fixed effect for the renal function group; Geometric mean ratio = 143.82, 90% CI 2-sided [118.306 to 174.848]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority or Other; ANOVA; The model includes fixed effect for the renal function group; Geometric mean ratio = 152.31, 90% CI 2-sided [125.287 to 185.166]

3. Primary Outcome: Maximum Concentration
Description: Maximum concentration of the analyte in plasma
Time Frame: as for outcome 2
Population: Treated patients
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
nmol/L | 1050 (19.1) | 984 (30.8) | 971 (26.2) | 990 (43.8)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Superiority or Other; ANOVA; The model includes fixed effect for the renal function group; Geometric mean ratio = 93.50, 90% CI 2-sided [72.236 to 121.015]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Superiority or Other; ANOVA; The model includes fixed effect for the renal function group; Geometric mean ratio = 92.18, 90% CI 2-sided [71.216 to 119.305]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Superiority or Other; ANOVA; The model includes fixed effect for the renal function group; Geometric mean ratio = 94.01, 90% CI 2-sided [72.630 to 121.674]

ADVERSE EVENTS:
Time Frame: From trial drug intake until the end-of-study examination visit, up to 12 days
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 2/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=8) | Mild Renal Impairment (N=8) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.